CLINICAL TRIAL: NCT03804203
Title: SHort Course Accelerated RadiatiON Therapy (SHARON) in Palliative Treatment of Esophageal Cancer: an Interventional, Randomized, Multicentric Study
Brief Title: Short Course Radiation Therapy in Palliative Treatment of Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT 15-07 SHARON ESOPHAGUS
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Cancer; Radiotherapy; Palliative Care
Keywords: Short Course Radiotherapy; Symptomatic esophageal lesions
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment (Active Comparator): patients in this group are treated with 3000 cGy in 10 daily fraction
  Interventions: Radiation: standard treatment
- short course treatment (Experimental): patients in this group are treated with 2000 cGy in 4 fractions administered twice a day (at least 6-8 hours interval)
  Interventions: Radiation: short course treatment

INTERVENTIONS:
Radiation: standard treatment — 3000 cGy in 10 daily fractions
  Arms: standard treatment
Radiation: short course treatment — 2000 cGy in 4 fractions administered twice a day
  Arms: short course treatment

SUMMARY:
Aim of the study is to assess efficacy of a short course radiation treatment in patients with symptomatic esophageal malignant lesions

DETAILED DESCRIPTION:
Standard treatment for esophageal lesions (3000 cGy in 10 daily fractions of 300 cGy each) is compared with experimental treatment (2000 cGy in 4 fractions of 500 cGy twice a day) to demonstrate non-inferiority of this scheme

ELIGIBILITY:
Inclusion Criteria:

* symptomatic esophageal malignant lesions (primary solid tumors or metastases from solid tumor);
* age>18 years;
* ECOG performance status 0-3
* no changes in supportive care in the week before radiotherapy

Exclusion Criteria:

* pregnancy
* previous irradiation of the same region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-11-08 (Estimated); Study Completion 2023-11-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of palliation using the short course scheme compared with the standard scheme: Likert scale | 3 months
  reduction of initial symptoms after radiotherapy, assessed with Likert scale (dysphagia, odynophagia, regurgitation, chest-back pain are evaluated as none-mild-moderate-severe)

SECONDARY OUTCOMES:
acute toxicity in the two treatment groups | 3 months
  incidence of treatment-related acute adverse events in the two arms of the study registered using Cooperative Group Common Toxicity Criteria
late toxicity in the two treatment groups | 12 months
  incidence of treatment-related adverse events in the two arms of the study registered using RTOG/EORTC Late Radiation Morbility Scoring Schema
Quality of Life (QoL): EORTC questionnaire C15-PAL | 12 months
  changes in QoL after the treatment assessed using European Organization for Research and Treatment of Cancer (EORTC) questionnaire C15-PAL (a specific questionnaire from EORTC developed to assess the quality of life of palliative cancer care patients)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Principal Investigator — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, Unversity of Bologna, S. Orsola-Malpighi Hospital
Locations (1):
- Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine- DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No